CLINICAL TRIAL: NCT06354894
Title: Riduzione e Sintesi Delle Fratture Del Terzo Prossimale d'Omero: Confronto Prospettico Tra Placca e Viti e Pinning Percutaneo
Brief Title: Percutaneous Pinning Versus Plate and Screws for Surgical Fixation of Proximal Humeral Fractures
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: MACOXS; 133/2020/U (Registry Identifier: MACOXS)
Record Dates: First submitted 2024-03-18; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Proximal Humeral Fractures
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients affected by proximal humeral fracture
  Interventions: Device: Proximal humeral fracture fixation

INTERVENTIONS:
Device: Proximal humeral fracture fixation — percutaneous pinning VS plate and screws

SUMMARY:
The aim of this multicenter nonrandomised study is to prospectively compare the clinical and radiographic results of two different techniques of surgical fixation of proximal humeral fractures: percutaneous pinning versus plate and screws.

ELIGIBILITY:
Inclusion Criteria:

* > 18 year old
* proximal humeral fracture
* both X-rays and CT scan available

Exclusion Criteria:

* dementia
* psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by proximal humeral fractures who consent to participate the study and whose fracture was considered to be treated with surgical fixation either with percutaneous pinning or with plate and screws
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score (OSS) | 1 year
  Patient reported outcome. Score from 0 to 48 points (with the higher score being the better)
Quick Disabilities of the arm, shoulder and hand (DASH) score | 1 year
  The questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms ranging from 0 (no disability) to 100 (most severe disability)
Subjective Shoulder Value (SSV) | 1 year
  The subjective shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder during ADLs (from 0% to 100%, with the higher score being the better)
Radiographic outcomes | 1 year
  Shoulder x-rays will be reviewed by a panel of experts in shoulder traumatology who will be asked to define the result as:
  * normal
  * nonunion
  * malunion
  * avascular necrosis
  * infection

CONTACTS AND LOCATIONS:
Locations (1):
- San Luigi Gonzaga Hospital, Orbassano, Turin, Italy